CLINICAL TRIAL: NCT02955316
Title: Irritable Bowel Syndrome Survey in Gastroenterological Adult Outpatients in China
Acronym: IRONS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1844R00004
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-10

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to estimate the overall prevalence of IBS medically diagnosed and diagnosed using Rome III or IV criteria in GI adult outpatients in China.

DETAILED DESCRIPTION:
This is a multicentre, nationwide and cross-sectional study carried out in China, covering 30 sites and 3000 patients totally. As for the ratio of tertiary to secondary general hospitals is approximately 1:4 in China, 6 tertiary and 24 secondary hospitals will be randomly selected in this study.To adapt the representativeness of the data with the operational feasibility, 30 tertiary and 120 secondary hospitals will be randomly selected over the 6 geographic regions (north, northeast, east, south central, southwest and northwest). Among those, 1 tertiary and 4 secondary hospitals in each region will be further selected based on GI department setup, willingness to participate in the study, capability and primary investigator's consideration. Within participated hospitals, subjects will be enrolled consecutively from all the outpatients of GI department to minimize selection bias. 3000 subjects will be allocated to tertiary and secondary hospitals with a ratio of 1:1. In general, 250 subjects will be enrolled from tertiary hospitals and 250 subjects will be enrolled from secondary hospitals for each region. During the subject enrolment, the investigator will firstly explain the purpose of the study to consecutive GI patients and written informed consents will be obtained. Then qualified patients will be given a questionnaire and finish it during waiting time. After receiving questionnaires, IBS diagnosis will be made by investigators based on Rome III or Rome IV IBS diagnostic criteria. Subjects will be identified as medically diagnosed with IBS if they have been diagnosed by their clinicians. And subjects will be classified as IBS sufferers without medical diagnosis if they satisfy Rome III or Rome IV diagnostic criteria and have not received IBS diagnosis from physicians. For IBS patients, either medically diagnosed or diagnosed with IBS criteria, investigators will collect all the information on demographic features, disease characteristics and current treatment status. For non-IBS patients, only demographic information will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of subject informed consent
2. Consecutive female and/or male GI outpatients aged 18 years and over

Exclusion Criteria:

1. Subject with a cognitive condition and unable to finish the questionnaire
2. Subject has an acute or chronic non-GI condition; e.g., doesn't record a 'yes' response to the question, 'Do you have a gut problem?'

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: gastroenterological adult outpatients
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
IBS prevalence in GI adult outpatients in China | one day
  Overall prevalence of IBS medically diagnosed and diagnosed using Rome III or IV criteria in GI adult outpatients in China.

SECONDARY OUTCOMES:
Overall and subgroups' prevalence of medically diagnosed IBS in GI adult outpatients | one day
  Overall prevalence and prevalence of IBS-C, D, M, U of medically diagnosed IBS adult outpatients.
Overall and subgroups' prevalence of IBS sufferers in GI adult patients without medical diagnosis | one day
  Overall prevalence and prevalence of IBS-C, D, M, U of IBS sufferers in GI adult patients without medical diagnosis
Identify demographic features of IBS and non-IBS outpatients | one day
  Demographic features of IBS and non-IBS outpatients: age, gender, occupation, use of smoking and alcohol, diet, sleeping habit
Identify disease characteristics of IBS outpatients | one day
  Disease characteristics of IBS outpatients: reason for visit to clinic, time of symptoms occur and diagnosis, previous diagnosis, bothersomeness of symptoms, frequency of symptoms, severity of symptoms, absence of work
Assess the current treatment status of IBS outpatients | one day
  Current treatment status: hospital visit frequency, previous medicine use, concomitant medications, treatment efficacy, treatment satisfaction, cost of therapy
Estimate the overall and subgroups' prevalence of IBS diagnosed by Rome III criteria in GI adult patients | one day
  Overall prevalence and prevalence of IBS-C,D,M,U of IBS diagnosed by Rome III criteria in GI adult outpatients in China
Estimate the overall and subgroups' prevalence of IBS diagnosed by Rome IV criteria in GI adult patients | one day
  Overall prevalence and prevalence of IBS-C,D,M,U of IBS diagnosed by Rome IV criteria in GI adult outpatients in China.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Hou, PhD, Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Research Site, Wuhan, Hubei, China

REFERENCES:
- See also: D1844R00004 CSR synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4419&filename=D1844R00004%20CSR%20synopsis.pdf